CLINICAL TRIAL: NCT02931500
Title: MachIne LEarning for Identification of Future Development of cardiovaScular and meTabOlic Disease: a NationwidE Time-series Cohort Study (MILESTONE)
Brief Title: Machine Learning for Identification of Future Disease Development: A Nationwide Cohort Study (MILESTONE)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hyuk-Jae Chang, Professor, Yonsei University
Other Study IDs: 4-2016-0383
Record Dates: First submitted 2016-07-21; First posted 2016-10-13 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Cardiovascular Disease; Metabolic Disease
Keywords: machine learning; cohort study
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To develop machine learning algorithms for the identification of future development of cardiovascular and metabolic disease

DETAILED DESCRIPTION:
The MILESTONE trial is retrospective and data review study with health checkup data from the National Health Insurance Services(NHIS) in Korea. The data will be included general health examination for individuals , type of health insurance, medical bill details, medical histories, treatment and prescriptions about 514,795 individuals who were over 40 years old.

ELIGIBILITY:
Inclusion Criteria:

* The Subject who is got health checkup between 2002 and 2013, and had been recorded the health checkup result to the National Health Insurance Service(NHIS) in South Korea.

Exclusion Criteria:

* Persons whose disease development is not identified from the records due to emigration or disappearance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data which is health checkup record about 510,000 Subjects between 2002 and 2013 from National Health Insurance Service (NHIS) in South Korea.
Sampling Method: Probability Sample
Enrollment: 510000 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy in prediction of development of cardiovascular and metabolic disease using machine learning algorithm | 6months

SECONDARY OUTCOMES:
Accuracy in prediction of development of cardiovascular and metabolic disease using logistic regression analysis | 6months
Accuracy in prediction of development of cardiovascular and metabolic disease using Framingham risk score | 6months

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk-Jae Chang, PhD, Principal Investigator — Yonsei Univerity
Locations (1):
- Yonsei University Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cho IJ, Sung JM, Kim HC, Lee SE, Chae MH, Kavousi M, Rueda-Ochoa OL, Ikram MA, Franco OH, Min JK, Chang HJ. Development and External Validation of a Deep Learning Algorithm for Prognostication of Cardiovascular Outcomes. Korean Circ J. 2020 Jan;50(1):72-84. doi: 10.4070/kcj.2019.0105. Epub 2019 Aug 19. PMID 31456363
- [Derived] Cho IJ, Sung JM, Chang HJ, Chung N, Kim HC. Incremental Value of Repeated Risk Factor Measurements for Cardiovascular Disease Prediction in Middle-Aged Korean Adults: Results From the NHIS-HEALS (National Health Insurance System-National Health Screening Cohort). Circ Cardiovasc Qual Outcomes. 2017 Nov;10(11):e004197. doi: 10.1161/CIRCOUTCOMES.117.004197. PMID 29150537